CLINICAL TRIAL: NCT05263076
Title: Uterine Transplantation and Pregnancy Induction in Women Affected by Absolute Uterine Factor Infertility
Brief Title: Uterine Transplant for Women With Absolute Uterine Factor Infertility (AUFI)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: John Goss (Other)
Responsible Party: Sponsor-Investigator, John Goss, Professor and Chief, Division of Abdominal Transplantation, Department of Surgery, Baylor College of Medicine
Organization: Baylor College of Medicine (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H-49601
Record Dates: First submitted 2022-01-18; First posted 2022-03-02 (Actual); Last update posted 2025-05-07 (Actual); Status verified 2025-05

CONDITIONS: Mayer Rokitansky Kuster Hauser Syndrome; Absence of Uterus; Infertility of Uterine Origin
Keywords: Uterine Transplant; AUFI; Absolute Uterine Factor Infertility; Infertility; MRKH
MeSH Terms: conditions — Mullerian aplasia; Infertility

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Uterine Transplant (Experimental): uterus transplantation from living or deceased donor.
  Interventions: Other: Uterine Transplant

INTERVENTIONS:
Other: Uterine Transplant — Transplant of a uterus from a live or deceased donor.

SUMMARY:
Absolute Uterine Factor Infertility (AUFI) is due to congenital or surgical absence of a uterus or the presence of a nonfunctional uterus. Until 2014, the only option for women affected by Absolute Uterine Factor Infertility (AUFI) was adoption or surrogate motherhood. Uterine transplant is a new form of transplant to treat AUFI. The technique of uterus transplant was developed in Sweden with the transplantation of the uterus from a living donor to a woman affected by AUFI. Approximately 80 uterine transplantations have been performed, more than 50 of which have occurred within the past 3 years. To date, 34 children have been born from mothers who have received a living donor uterine transplant.

This is a prospective study to treat Absolute Uterine Factor Infertility (AUFI) through uterine transplantation utilizing a uterus from a living or deceased donor resulting in live birth. A total of 10 biologically female (XX Karyotype) subjects will receive a uterine transplant.

DETAILED DESCRIPTION:
BACKGROUND: The feasibility of uterine transplant has been studied for more than a decade. The clinical concept and the technical aspects were first tested and proven in non-primates and then in primate experiments. In 2013, the first human trial started at the University of Gothenburg in Sweden. In 2014, the first live birth from a woman who had received a uterine transplant was announced (1). This first live birth was then followed by additional births. Uterine transplant may provide an additional option for women with Absolute Uterine Factor Infertility (AUFI).

STUDY DESIGN: This trial will be conducted at Texas Children's Hospital - Pavilion for Women. Texas Children's Hospital was established in 1954. Today it has one of the nation's top pediatric transplant programs. The transplant center has performed more than 2000 solid organ transplants including liver, kidney, heart and lung transplants. This is a non-randomized, interventional study with the goal of achieving pregnancy and live birth of a child following uterine transplantation using either a live or deceased uterus donor. The investigators plan to perform 10 uterine transplants in this study.

The evaluation for receiving a uterine transplant will include consults with specialists and a variety of procedures. The consultations, tests and procedures will evaluate if the recipient is physically, emotionally, and mentally prepared to participate. After the evaluations are complete, the principal investigator and coordinator will present the findings to the rest of the uterine team. The team will decide if the subject is a candidate for moving forward to the IVF part of the screening process. After successful completion of egg retrieval and fertilization, the embryos will be banked. Only those study subjects that have four or more high quality embryos will be the criteria to be listed as uterine transplant recipients. Preimplantation Genetic Testing for Aneuploidy will be done. Once the subject has undergone uterine transplantation, she will be monitored for infection, rejection and other complications.

Once it has been determined that the study subject is ready for the embryo transfer, the subject will undergo a process to prepare the uterus to receive the embryo (embryo transfer). The endometrium will be stimulated to grow with estrogen until a desired thickness of the lining has been obtained. A second hormone, progesterone, will be given by injection daily until the endometrial lining is receptive to transfer of the embryo. On the day of the transfer, the embryo will be thawed and then transferred into the uterus by means of a sterile catheter system under ultrasound guidance to determine the proper placement of the embryo into the uterus. The study subject will be awake during this process. Twelve days later, blood tests will be performed to detect the pregnancy hormone, HCG. The levels of the pregnancy hormone and the estrogen and progesterone levels will be closely monitored. At eight weeks gestation, the study subject will undergo an ultrasound evaluation to see if there is viable pregnancy. The study subject will then be closely monitored by the fertility specialist until about 11 weeks, and then by a Maternal-Fetal Medicine (MFM) specialist.

All deliveries will be performed via cesarean section. Following delivery, the subject will have the opportunity to discuss with the transplant and Ob/Gyn team the possibility of a second pregnancy or explant of the uterus. If a second pregnancy is anticipated the subject must be deemed medically stable to undergo the embryo transfer and a second-high risk pregnancy. The subject and team will determine the timeline for a second pregnancy if the subject so chooses. If the subject chooses to undergo a second pregnancy, she will be followed by a Maternal Fetal Medicine specialist and delivery via repeat cesarean delivery. After delivery of the first pregnancy, a decision about a second pregnancy or an explant will not be made until at least 60 days post-delivery to allow time to evaluate the health of the newborn as well as the candidacy of the subject for a possible second pregnancy (if desired). In the case of a second pregnancy, the plan will be to perform a hysterectomy of the uterine allograft at the time of cesarean delivery of the second child.

The transplanted uterus will be from either living or deceased donors. TXTC wants to be certain that the living donor's decision to donate is made freely, and with all of the information needed to consider donation. For that reason, TXTC has an agreement with the Living Bank that will serve as an independent third party advocating for the rights and needs of the donor through the evaluation and donation process. UNOS is the only source for deceased donor organs. Locally, TXTC works with the Lifegift OPO to procure organs for transplant.

ELIGIBILITY:
RECIPIENT INCLUSION CRITERIA

1. Women who are diagnosed with Absolute Uterine Factor Infertility (AUFI) and who have at least one functioning ovary.
2. Women of childbearing age (20-40 years old) who are biologically female (XX karyotype).
3. Subjects will not have active human 142 papillomavirus (HPV) or active cervical dysplasia present.
4. Subjects will have negative testing for Gonorrhea Chlamydia and Syphilis and will not have any active bacterial vaginosis or candida infection. (Subjects with previously treated STDs will be included if the infection is no longer present and has no impact. If a subject develops an STD/infection pre-operatively, she will be treated and monitored for a period of 3 months until she is no longer affected. She will then become eligible for transplant. If a subject develops an STD/infection after transplant/during pregnancy she will be treated appropriately. Prior to the embryo transfer the patient will be tested and treated if necessary. Any patient with an active STD/infection will be ineligible for any elective procedure until she is tested and treated appropriately.)
5. Subjects who are HSV-2 negative or who have a history of HSV-2 with no current symptoms. Subjects may require preventative maintenance per study doctor discretion.
6. Subjects have received counseling regarding all fertility options and alternatives to uterine transplant such as adoption or surrogate pregnancy.
7. Subjects are willing to undergo in-vitro fertilization to obtain the necessary 4 viable embryos required for eligibility for transplant if they have not already banked 4 viable embryos.
8. Subjects have been evaluated by a fertility specialist and determined to have good ovarian reserve and reproductive potential.
9. Subjects must agree that in the event of withdrawal from the study while the transplanted uterus is in place, unless she is enrolled in an equivalent uterine transplant program, she will be required to undergo a hysterectomy for her own safety.
10. Subject meets psychological recipient criteria.
11. Subject must be willing to complete questionnaires about their infant's growth and development and return them to the study team.

RECIPIENT EXCLUSION CRITERIA

1. Subject with Diabetes Mellitus Type I and II by medical history or elevated hemoglobin A1c blood test.
2. Subject has known hypersensitivity to Tacrolimus, Thymoglobulin or Everolimus.
3. Subject with a diagnosis of hypertension, or any other significant medical condition that makes this procedure unsafe or is a contraindication to surgery or anesthesia.
4. Subject who has a history of solid organ or bone marrow transplant, per investigator's discretion.
5. Subject who has a history of cancer, per investigator's discretion.
6. Subject with a body mass index >30.
7. Subject with an active infection including candida and/or bacterial vaginosis.
8. Subject who is seropositive for HIV, HBV, HCV.
9. Subject with technical obstacles as per anatomical malformations, which pose a high surgical risk in the judgment of the investigator.
10. Subject unwilling or unable to comply with study requirements.
11. Subject unable to undergo in-vitro fertilization or not cleared for transplant.
12. Subject who has smoked within the last 6 months.
13. Subject who has alcohol or drug abuse within 12 months of screening.
14. Subject with any pre-existing clinical or medical conditions that would put the subject at an increased risk. Of note, for Mayer-Rokitansky-Kuster-Hauser (MRKH) syndrome, the investigators will favor Type 1 variants as Type 2 is associated with skeletal/spinal and renal anomalies, making them higher risk candidates.

DONOR INCLUSION CRITERIA

1. Women must be between 25-65 years of age. If a subject is less than 40 years old she must be certain that she does not wish to carry more children, and she will attest to this decision.
2. Subjects will not have active human 142 papillomavirus (HPV) or active cervical dysplasia present.
3. Subjects will have negative testing for Gonorrhea, Chlamydia and Syphilis and will not have any active bacterial vaginosis or candida infection. (Subjects with previously treated STDs will be included if the infection is no longer present and has no impact. If a subject develops an STD/infection pre-operatively, she will be treated and monitored for a period of 3 months until she is no longer affected. Any patient with an active STD/infection will be ineligible for any elective procedure until she is tested and treated appropriately.)
4. Subjects who are HSV-2 negative, or have a history of HSV-2 but with no current symptoms. Subjects may require preventative maintenance per study doctor discretion.
5. Subjects will have a normal uterus on sonogram and CT.
6. Subjects will have normal psychological donor criteria (if living).
7. Subjects will have had at least one prior full term live birth.

DONOR EXCLUSION CRITERIA

1. Donor over the age of 65.
2. Body mass index >30.
3. Subject with an active infection including candida and/or bacterial vaginosis.
4. Subject who is seropositive for HIV, HBV, HCV
5. Subject who has had cancer in the last five years.
6. Subject with any pre-existing clinical or medical condition that would place the subject at an increased risk or would be a contraindication to surgery or anesthesia.
7. Subject who has smoked within the last 6 months.
8. Subject who has alcohol or drug abuse within 12 months of screening.
9. Subject unwilling or unable to comply with study requirements.

Ages: 20 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2022-06-03 (Actual); Primary Completion 2030-12 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
Number of participants that have successful procurement of a viable uterus for transplant. | Day of organ procurement immediately post-operative
  A viable uterus is a uterine allograft that is fully procured and is suitable for transplantation into the recipient. This is measured at the time of procurement by visible inspection to ensure the vascular structures (uterine artery and vein) are not injured and the vaginal cuff is intact.
Number of participants that have a score of II or less on the Clavian-Dindo Scale. | 30 days post-operative
  Each patient will be reviewed and any complications scored using the Clavian Dindo Scale.
Successful transplantation of a human uterus with achievement of menstrual cycles | 3 months post-operative
  As determined by 1. Achievement of menstrual cycles at 3 months post-operative, and 2. Graft viability measured by assessing blood flow via ultrasound and using cervical biopsies to look for ischemia or allograft rejection.
Successful establishment of a pregnancy via in vitro fertilization | 6 weeks post IVF
  Visibility of a gestational sac on US at 6 weeks
Successful live birth | at birth
  Viable infant born ≥ 23 weeks gestation

CONTACTS AND LOCATIONS:
Overall Officials: John Goss, M.D., Principal Investigator — Baylor College of Medicine
Locations (1):
- Texas Children's Hospital, Houston, Texas, United States